CLINICAL TRIAL: NCT01490281
Title: Land- and Water-Based Exercise Intervention in Women With Fibromyalgia: The Al-Andalus Physical Activity Randomised Control Trial
Brief Title: Exercise in Women With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Co-Coordinator, Junior Research Fellow, Universidad de Granada
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: DEP2010-15639; CTCD-201000019242-TRA (Other Grant/Funding Number: CTCD-201000019242-TRA)
Record Dates: First submitted 2011-12-05; First posted 2011-12-12 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; exercise; physical activity; pain
MeSH Terms: conditions — Fibromyalgia; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- water-based exercise intervention (Experimental)
  Interventions: Behavioral: water-based exercise
- land-based exercise intervention (Experimental)
  Interventions: Behavioral: land-based exercise intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: water-based exercise — Interventions will consist of aerobic, muscular strength and flexibility exercises in the water
  Arms: water-based exercise intervention
Behavioral: land-based exercise intervention — Interventions will consist of aerobic, muscular strength and flexibility exercises in the land
  Arms: land-based exercise intervention

SUMMARY:
Background The Al-Andalus physical activity intervention study is a randomised control trial to investigate the effectiveness of a land- and water-based exercise intervention for reducing the overall impact of fibromyalgia (primary outcome), and for improving tenderness and pain-related measures, body composition, functional capacity, physical activity and sedentary behaviour, fatigue, sleep quality, health-related quality of life, and cognitive function (secondary outcomes) in women with fibromyalgia.

Methods One hundred eighty women with fibromyalgia (age range: 35-65 years) will be recruited from local associations of fibromyalgia patients in Andalucía (Southern Spain). Patients will be randomly assigned to a usual care (control) group (n=60), a water-based exercise intervention group (n=60) or a land-based exercise intervention group (n=60). Participants in the usual care group will receive general physical activity guidelines and participants allocated in the intervention groups will attend three non-consecutive training sessions (60 minutes each) per week during 24 weeks. Both exercise interventions will consist of aerobic, muscular strength and flexibility exercises.

Discussion The investigators study attempts to reduce the impact of fibromyalgia and improve patients' health status by implementing two types of exercise interventions. Results from this study will help to assess the efficacy of exercise interventions for the treatment of fibromyalgia. If the interventions would be effective, this study will provide low-cost and feasible alternatives for health professionals in the management of fibromyalgia. Results from the Al-Andalus physical activity intervention will help to better understand the potential of regular physical activity for improving the well-being of women with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-65 years.
* Meeting the American College of Rheumatology criteria: widespread pain for more than 3 months, and pain with 4 kg/cm of pressure reported for 11 or more of 18 tender points.
* Not to have other severe somatic or psychiatric disorders, or other diseases that prevent physical loading (Answer "no" to all questions on the Physical Activity Readiness Questionnaire-PAR-Q ).
* Not to be engaged in regular physical activity >20 minutes on >3 days/week.
* Planning to stay in the same Association during the study.
* Able to ambulate, with or without assistance.
* Able to communicate.
* Informed consent: Must be capable and willing to provide consent.

Exclusion Criteria:

* Acute or terminal illness.
* Myocardial infarction in the past 3 months.
* Not capable to ambulate.
* Unstable cardiovascular disease or other medical condition.
* Upper or lower extremity fracture in the past 3 months.
* Severe dementia (MMSE<10).
* Unwillingness to either complete the study requirements or to be randomised into control or training group.
* Presence of neuromuscular disease or drugs affecting neuromuscular function.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall impact of fibromyalgia | Participants will be followed over 24 weeks
  The primary outcome will be assessed with the fibromyalgia Impact Questionnaire (FIQ). FIQ is a self-administered questionnaire, comprising 10 subscales of disabilities and symptoms (physical function, work missed day, job ability, feel good, pain, fatigue, sleep, stiffness, anxiety and depression) and has been validated for Spanish fibromyalgia patients. The total scores range from 0 to 100, with a higher score indicating greater effect of the condition on the person's life.

SECONDARY OUTCOMES:
Tenderness | Participants will be followed over 24 weeks
  A total of 18 tender points will be assessed according to the American College of Rheumatology criteria for classification of fibromyalgia using a standard pressure algometer (FPK 20; Effegi, Alfonsine, Italy). The tender point count, total count of positive tender points, will be recorded for each participant. The algometer score will be calculated as the sum of the minimum pain-pressure values obtained for each tender point.
Visual analogic scale for pain | Participants will be followed over 24 weeks
  Visual analogic scale for pain. This is a simple assessment tool consisting of a 10 cm line with 0 on one end, representing no pain, and 10 on the other, representing the worst pain ever experienced, which a patient marks to indicate the severity of her pain in the present moment. This scale will also be administered before and after each session during the intervention, to assess the acute effect of exercise on pain.
The Pain Catastrophizing Scale | Participants will be followed over 24 weeks
  It assesses three factors: rumination, magnification and helplessness associated to pain. It includes 13 items measured on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time). Higher scores indicate a greater tendency to catastrophize pain symptoms.
Body composition | Participants will be followed over 24 weeks
  Weight and height will be measured, body mass index [weight (kg)/height(m2)] will be calculated, and skeletal muscle mass, total body water and fat free mass will be estimated with bioelectrical impedance analysis (InBody R20; Biospace, Gateshead, UK).
Functional capacity | Participants will be followed over 24 weeks
  Participants' functional capacity will be assessed by field-based fitness tests following the standardised Functional Senior Fitness Test Battery
Fatigue | Participants will be followed over 24 weeks
  The Multidimensional Fatigue Inventory will be used to measure fatigue severity, and comprises five subscales: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation.
Sleep Quality | Participants will be followed over 24 weeks
  Pittsburgh Sleep Quality Index will be used to assess sleep quality and disturbances
Health-related quality of life | Participants will be followed over 24 weeks
  We will determine patients' quality of life with the Short-Form Health Survey 36 (SF-36)
Cognitive function | Participants will be followed over 24 weeks
  The Mini Mental State Examination (MMSE) will be used to evaluate cognitive capacity and severity of dementia for the exclusion criteria

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Granada, Spain

REFERENCES:
- [Derived] Carbonell-Baeza A, Ruiz JR, Aparicio VA, Ortega FB, Munguia-Izquierdo D, Alvarez-Gallardo IC, Segura-Jimenez V, Camiletti-Moiron D, Romero A, Estevez-Lopez F, Samos B, Casimiro AJ, Sierra A, Latorre PA, Pulido-Martos M, Femia P, Perez-Lopez IJ, Chillon P, Girela-Rejon MJ, Tercedor P, Lucia A, Delgado-Fernandez M. Land- and water-based exercise intervention in women with fibromyalgia: the al-Andalus physical activity randomised controlled trial. BMC Musculoskelet Disord. 2012 Feb 15;13:18. doi: 10.1186/1471-2474-13-18. PMID 22336292